CLINICAL TRIAL: NCT05377229
Title: MarginProbe 2.0 Data Collection Protocol
Status: Completed | Type: Observational
Sponsor: Dilon Medical Technologies Ltd. (Industry)
Responsible Party: Sponsor
Organization: Dilon Technologies Inc. (Industry)
Other Study IDs: CP-13-001
Record Dates: First submitted 2022-05-09; First posted 2022-05-17 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer
Keywords: MarginProbe; Breast Cancer; Lumpectomy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

INTERVENTIONS:
Device: MarginProbe2.0 — The MarginProbe System is an adjunctive diagnostic tool for identification of cancerous tissue at the margins of the ex-vivo lumpectomy specimen following primary excision and is indicated for intraoperative use, in conjunction with standard methods (such as intraoperative imaging and palpation) in patients undergoing breast lumpectomy surgery for previously diagnosed breast cancer.
  Other Names: MP2.0

SUMMARY:
Previous clinical studies with the MarginProbe (MP) system demonstrated the MP System diagnostic accuracy for identification of cancerous/abnormal tissue at the margins (≤ 1mm) of the ex-vivo lumpectomy specimen. The current study is a prospective data collection study with the enhanced technology, the MP2.0 System and is aimed at collecting data to optimize the system algorithm/procedure and to subsequently validate the system to demonstrate non-inferiority to the MP1.x system.

In this study, MP2.0 system will be used on ex-vivo lumpectomy specimens at the Operating Room (OR). The study will collect a library of case information data using the MP2.0 system in sequential cohorts of a minimum of 50 subjects until the software and procedure are optimized. The final analysis sample size will be determined and outlined in the SAP based upon the results of the optimization stage.

ELIGIBILITY:
Inclusion Criteria:

1. Women over 18 years of age
2. Diagnosed with cancer, undergoing lumpectomy or partial mastectomy procedure
3. Signed Informed Consent Form

Exclusion Criteria:

1. Undergoing re-excision procedure
2. Concurrent infectious disease
3. Pregnancy
4. Lactation
5. Previous surgery in the same site including open biopsy procedure, previous breast reduction or mastopexy in the operated breast
6. Prior radiation treatment in the operated breast
7. Participating in any other investigational study for either drug or device which can influence collection of valid data under this study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include measurements in cohorts of a minimum of 50 subjects up to a maximum of 1000 cases from women, aged 18 and above, undergoing breast lumpectomy/partial mastectomy surgery for previously diagnosed breast cancer.
Sampling Method: Probability Sample
Enrollment: 398 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2024-08-23 (Actual); Study Completion 2025-01-12 (Actual)

PRIMARY OUTCOMES:
Adverse Events (AEs) and Serious Adverse Events (SAEs) | During the lumpectomy surgery
  Adverse Events (AEs) and Serious Adverse Events (SAEs)
Collect MP2.0 data in cohorts of a minimum of 50 subjects to optimize MP2.0 algorithm and procedure. | During the lumpectomy surgery
  The cohorts will continue to be collected until a final algorithm is established and the cohort(s) can be collected with the final algorithm to determine the sensitivity and specificity to demonstrate non-inferiority to the MP1.x system.

CONTACTS AND LOCATIONS:
Locations (9):
- United States (8):
  - Glendale Adventist Medical Center, Glendale, California
  - Mercy Medical Center, Cedar Rapids, Iowa
  - Logan Health Breast Center, Kalispell, Montana
  - Englewood Health, Englewood, New Jersey
  - Health and Hospitals Corporation/Kings County, Brooklyn, New York
  - Northwell Northern Westchester, Mount Kisco, New York
  - Northwell Health, Staten Island, New York
  - Lehigh Valley, Bethlehem, Pennsylvania
- Hadassah Medical Organization, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No